CLINICAL TRIAL: NCT03995550
Title: A Randomised, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LEO 142397 in Healthy Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics After Single and Multiple Doses of LEO 142397 in Healthy People, Including Japanese
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Portfolio proritisation
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LP0184-1415; 2018-004470-10 (EudraCT Number)
Record Dates: First submitted 2019-06-21; First posted 2019-06-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2019-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Single ascending dose Cohort A (Experimental): Single dose of LEO 142397 or placebo.
  Interventions: Drug: LEO 142397; Drug: Placebo
- Single ascending dose Cohort B (Experimental): Single dose of LEO 142397 or placebo.
  Interventions: Drug: LEO 142397; Drug: Placebo
- Single ascending dose Cohort C (Experimental): 2 single doses, separated by a washout of ≥7 days.
  Interventions: Drug: LEO 142397; Drug: Placebo
- Single ascending dose Cohort D (Experimental): 2 single doses, separated by a washout of ≥7 days.
  Interventions: Drug: LEO 142397; Drug: Placebo
- Single ascending dose Cohort E (Experimental): Single dose of LEO 142397 or placebo.
  Interventions: Drug: LEO 142397; Drug: Placebo
- Single ascending dose Cohort F (Experimental): Single dose of LEO 142397 or placebo.
  Interventions: Drug: LEO 142397; Drug: Placebo
- Single ascending dose Cohort G (Experimental): Single dose of LEO 142397 or placebo.
  Interventions: Drug: LEO 142397; Drug: Placebo
- Single ascending dose Cohort H (Experimental): Single dose of LEO 142397 or placebo - tentative, female-only cohort (to be included only if the number of women recruited in the remaining cohorts is insufficient to assess the pharmacokinetics of LEO 142397 in women). Dose level ≥ that in Cohort C and ≤ that in Cohort D.
  Interventions: Drug: LEO 142397; Drug: Placebo
- Multiple ascending dose Cohort K (Experimental): Multiple doses of LEO 142397 or placebo.
  Interventions: Drug: LEO 142397; Drug: Placebo
- Multiple ascending dose Cohort L (Experimental): Multiple doses of LEO 142397 or placebo.
  Interventions: Drug: LEO 142397; Drug: Placebo
- Multiple ascending dose Cohort M (Experimental): Multiple doses of LEO 142397 or placebo.
  Interventions: Drug: LEO 142397; Drug: Placebo
- Multiple ascending dose Cohort N (Experimental): Multiple doses of LEO 142397 or placebo.
  Interventions: Drug: LEO 142397; Drug: Placebo
- Multiple ascending dose Cohort O (Experimental): Multiple doses of LEO 142397 or placebo.
  Interventions: Drug: LEO 142397; Drug: Placebo
- Multiple ascending dose Cohort P (Experimental): Multiple doses of LEO 142397 or placebo in Japanese-only subjects. Same dose level as for Cohort M.
  Interventions: Drug: LEO 142397; Drug: Placebo

INTERVENTIONS:
Drug: LEO 142397 — A compound in development by LEO Pharma A/S
Drug: Placebo — Placebo

SUMMARY:
This is the first clinical trial with LEO 142397. The purpose of the trial is to assess the safety and tolerability of LEO 142397, along with the pharmacokinetics (what the body does to the drug) and the pharmacodynamics (what the drug does to the body) in healthy people.

The trial consists of 2 parts:

* In Part 1, participants will receive a single dose of LEO 142397. There will be up to 8 different dose groups.
* In Part 2, participants will receive a daily dose of LEO 142397 for 14 days. There will be up to 6 different dose groups.

Each participant will be enrolled into 1 dose group in either Part 1 or Part 2.

ELIGIBILITY:
Key inclusion Criteria:

* Body mass index of 18.0-32.0 kg/m2, inclusive.
* In good health at screening and check-in as judged by the investigator based on medical history, physical examination, vital signs assessment, 12-lead electrocardiogram, and clinical laboratory evaluations:

  * Aspartate aminotransferase and alanine aminotransferase values ≤1.5 times the upper limit of normal.
  * Congenital nonhaemolytic hyperbilirubinaemia (including suspicion of Gilbert's syndrome) is not acceptable.
  * Haemoglobin value, neutrophil count, and lymphocyte count ≥ the lower limit of normal.
* Female subjects of childbearing potential must use a highly effective form of birth control, in conjunction with adequate barrier contraception, from randomisation until 90 days after the follow-up visit.
* Male subjects with female partner of childbearing potential must use adequate male barrier contraception, in conjunction with a highly effective form of female contraception for the partner, from randomisation until 90 days after the follow-up visit.

Key exclusion criteria:

* Any surgical or medical condition that might significantly alter the absorption, distribution, metabolism, or excretion of any drug.
* Any medication, including St. John's wort, known to chronically alter drug absorption or elimination processes within 30 days prior to the first dose.
* History of any significant infectious disease, as assessed by the investigator, within 2 weeks prior to the first dose.
* Current active tuberculosis based on QuantiFERON-TB Gold test.
* Positive hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus antibodies at screening.
* Electrocardiogram abnormalities at screening or check-in.
* Smoking of >10 cigarettes per day, on average, within the last 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Part 1. Number of treatment-emergent adverse events per subject | From Day 1 (postdose) up to Day 8
Part 1. Having clinically significant abnormalities in systolic blood pressure | From Day 1 (postdose) up to Day 8
  Clinical significance (yes/no) of abnormal values as judged by the investigator
Part 1. Having clinically significant abnormalities in diastolic blood pressure | From Day 1 (postdose) up to Day 8
  Clinical significance (yes/no) of abnormal values as judged by the investigator
Part 1. Having clinically significant abnormalities in heart rate | From Day 1 (postdose) up to Day 8
  Clinical significance (yes/no) of abnormal values as judged by the investigator
Part 1. Having clinically significant abnormalities in oral body temperature | From Day 1 (postdose) up to Day 8
  Clinical significance (yes/no) of abnormal values as judged by the investigator
Part 1. Having an abnormal ECG | From Day 1 (postdose) up to Day 8
  ECG: electrocardiogram. Abnormal ECG (yes/no) defined as: QT interval corrected for heart rate using Fridericia's formula (QTcF) of >450 msec for males / >470 msec for females, or change from baseline of >30 msec
Part 2. Number of treatment-emergent adverse events per subject | From Day 1 (postdose) up to Day 21
Part 2. Having clinically significant abnormalities in systolic blood pressure | From Day 1 (postdose) up to Day 21
  Clinical significance (yes/no) of abnormal values as judged by the investigator
Part 2. Having clinically significant abnormalities in diastolic blood pressure | From Day 1 (postdose) up to Day 21
  Clinical significance (yes/no) of abnormal values as judged by the investigator
Part 2. Having clinically significant abnormalities in heart rate | From Day 1 (postdose) up to Day 21
  Clinical significance (yes/no) of abnormal values as judged by the investigator
Part 2. Having clinically significant abnormalities in oral body temperature | From Day 1 (postdose) up to Day 21
  Clinical significance (yes/no) of abnormal values as judged by the investigator
Part 2. Having an abnormal ECG | From Day 1 (postdose) up to Day 21
  ECG: electrocardiogram. Abnormal ECG (yes/no) defined as: QT interval corrected for heart rate using Fridericia's formula (QTcF) of >450 msec for males / >470 msec for females, or maximum change from baseline of >30 msec

SECONDARY OUTCOMES:
Part 1. AUC0-∞ | Derived from plasma concentration-time profile from 0-48 hours postdose
  AUC0-∞: area under the plasma concentration-time curve from time zero to infinity
Part 1. Cmax | Derived from plasma concentration-time profile from 0-48 hours postdose
  Cmax: maximum plasma concentration
Part 2. Accumulation ratio | Derived from plasma concentration-time profile from 0-24 hours postdose on Day 1 and Day 14
Part 2. AUC0-24 | Derived from plasma concentration-time profile from 0-24 hours postdose on Day 1 and Day 14
  AUC0-24: area under the plasma concentration-time curve from time zero to 24 hours postdose
Part 2. Cmax | Derived from plasma concentration-time profile from 0-24 hours postdose on Day 1 and Day 14
  Cmax: maximum plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (1):
- Covance Clinical Research Unit Ltd., Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes